CLINICAL TRIAL: NCT01977443
Title: Evaluation of the Therapeutic Efficacy of APD-209 Eye Drops in Treatment of Acute Phase Adenoviral-Induced Epidemic Keratoconjunctivitis (EKC). A Randomised, Double-Masked, Placebo-Controlled, Multi-Centre Proof-of-Concept Study
Brief Title: Therapeutic Efficacy of APD-209 Eye Drops in Treatment of Epidemic Keratoconjunctivitis (EKC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adenovir Pharma AB (Industry)
Collaborators: TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012/ADE002; 2012-005694-31 (EudraCT Number)
Record Dates: First submitted 2013-10-31; First posted 2013-11-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Viral Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Viral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APD-209 Eye drops (Active Comparator): APD-209 Eye drops
  Interventions: Drug: APD-209 Eye drops
- APD-209 Placebo Eye drops (Placebo Comparator): APD-209 Placebo Eye drops
  Interventions: Drug: APD-209 Placebo Eye drops

INTERVENTIONS:
Drug: APD-209 Eye drops
  Arms: APD-209 Eye drops
Drug: APD-209 Placebo Eye drops
  Arms: APD-209 Placebo Eye drops

SUMMARY:
A randomized, double-masked, placebo-controlled, multi-centre phase IIa proof-of-concept study to evaluate efficacy and safety of APD-209 Eye drops for treatment of acute phase adenovirus-induced EKC. The aims of the study are to investigate the therapeutic efficacy of APD-209 Eye drops as measured by adenoviral load, time to viral eradication, clinical resolution of EKC (objective and subjective assessments), presence of opacities, visual acuity and frequency of second eye infections, and to assess the safety and tolerability of APD-209 Eye drops in EKC infected eyes.

ELIGIBILITY:
Inclusion Criteria:

The patients have to meet all of the following criteria to be eligible to enter the study:

* Willing and able to provide informed consent.
* Men or women aged 18 years or above with onset of adenoviral EKC symptoms in at least one eye, as clinically diagnosed and with symptoms appearing within less 7 days at the time of giving informed consent.
* Using adequate contraceptive measures

Exclusion Criteria:

* Known or suspected allergy to any ingredient of the IMP or placebo.
* Symptoms correlating with EKC since more than 7 days.
* Diagnosis of other significant disease(s) than EKC in the eye.
* Diagnosis of bacterial or fungal ocular infections.
* Use of antibiotics or corticosteroids by any route (except intravitreal corticosteroids) within 14 days prior to inclusion. Ocular antibiotics may, however, be used until 2 hours prior to first dose of IMP, but are thereafter prohibited during the study.
* Use of immunosuppressive medications (including intravitreal corticosteroids) within 6 months prior to inclusion.
* Use of antiviral medications within 7 days prior to inclusion.
* Usage of any medication or herbal medicinal product with documented adverse reactions affecting the eyes.
* Usage of any medication or herbal medicinal product for ocular administration at inclusion.
* Female patients: currently pregnant or breast-feeding or intending to become pregnant during the study period.
* Known or suspected drug abuse.
* Usage of contact lenses during the study.
* Participation in any other interventional clinical study within 30 days prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the adenoviral load in epidemic keratokonjunctivitis (EKC) infected eyes following topical treatment with APD-209 Eye drops compared to placebo. | 14 days
  Viral load in tear liquid from EKC infected eyes, as measured by the area under the curve (AUC) at 3-14 days from start of treatment.

SECONDARY OUTCOMES:
Assess the time to viral eradication in EKC infected eyes following treatment with APD-209 Eye drops compared to placebo. | 14 days
  The time point of viral eradication in tear liquid from EKC infected eyes, defined as the time Point when viral load=0 or below the lower limit of quantification (LLOQ).
Evaluate the effect of APD-209 Eye drops on clinical resolution of EKC, as measured by objective and subjective assessment of scaled clinical symptoms, compared to placebo. | 14 days
  Resolution of acute ocular symptoms at each time of assessment, as measured by objective (Investigator-based) assessment of conjunctival discharge and redness.
Evaluate the presence of opacities (quantitatively and qualitatively) following treatment with APD-209 Eye drops compared to placebo. | 14 days
  Presence and location of opacities at each time of assessment, as measured by slit lamp examination.
Assess the visual acuity following treatment with APD-209 Eye drops compared to placebo. | 28 days
  Visual acuity at each time of assessment by use of the logarithm of the Minimum Angle of Resolution (LogMAR) chart.
Assess the frequency of second eye infections. | 14 days
  Occurrence of second eye infection.
Assess the safety and tolerability of APD-209 Eye drops. | 14 days
  Safety variables: adverse events (AEs) (nature and incidence), Physical examination, vital signs, laboratory safety assessments (haematology, clinical chemistry and urinalysis)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Gustaf Laurell, MD PhD, Principal Investigator — St Eriks Eye Hospital
Locations (10):
- Germany (7):
  - Augenklinik Universitätzmedizin Charité, Berlin
  - Augenklinik Köln, Merheim, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitäts-Augenklinik Freiburg, Freiburg im Breisgau
  - Universitäts-klinikum Schleswig-Holstein, Lübeck
  - Augenklinik, Universitätsklinikum Tübingen, Tübingen
  - Universitäts-Augenklinik, Würzburg
- Poland (2):
  - Katowice University Hospital, Katowice
  - P. Oleksy Centrum Medyczne Uno-Med, Tarnów
- St Eriks Eye Hospital, Stockholm, Sweden